CLINICAL TRIAL: NCT02891447
Title: A Phase II Study of Cytoreduction, Gastrectomy, and Hyperthermic Intraperitoneal Chemoperfusion (HIPEC) in Patients With Gastric Adenocarcinoma and Carcinomatosis or Positive Cytology
Brief Title: Heated Mitomycin and Cisplatin During Surgery in Treating Patients With Stomach or Gastroesophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0269; NCI-2018-02341 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0269 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Hyperthermic Intraperitoneal Chemotherapy; Mitomycin; Mitozytrex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (mitomycin, cisplatin) (Experimental): Patients undergo HIPEC comprised of mitomycin and cisplatin given intraperitoneally over 60 minutes during standard of care cytoreduction and gastrectomy.
  Interventions: Drug: Cisplatin; Drug: Hyperthermic Intraperitoneal Chemotherapy; Drug: Mitomycin

INTERVENTIONS:
Drug: Cisplatin — Given intraperitoneally
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Hyperthermic Intraperitoneal Chemotherapy — Undergo HIPEC
  Other Names: HIPEC
Drug: Mitomycin — Given intraperitoneally
  Other Names: Ametycine; MITO; MITO-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706

SUMMARY:
This phase II trial studies how well heated mitomycin and cisplatin during surgery work in treating patients with stomach or gastroesophageal cancer. Drugs used in chemotherapy, such as mitomycin and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Heating a chemotherapy solution and infusing it directly into the abdomen may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess overall survival from the date of diagnosis in subjects with stage IV gastric or gastroesophageal cancer and positive cytology or carcinomatosis after cytoreduction, gastrectomy, and hyperthermic intraperitoneal chemotherapy administration.

SECONDARY OBJECTIVES:

I. To assess the safety of cytoreduction, gastrectomy, and hyperthermic intraperitoneal chemotherapy administration for subjects with gastric or gastroesophageal cancer and positive cytology or carcinomatosis.

OUTLINE:

Patients undergo hyperthermic intraperitoneal chemotherapy (HIPEC) comprised of mitomycin and cisplatin given intraperitoneally over 60 minutes during standard of care cytoreduction and gastrectomy.

After completion of study treatment, patients are followed up within 4 weeks, and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Cytologic or histologic proof of adenocarcinoma of the stomach or gastroesophageal junction
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 60,000/Ul
* Serum creatinine =< 1.5 mg/dL
* Distant metastatic disease of peritoneum may be visualized on imaging:

  * Positive peritoneal cytology
  * Carcinomatosis on diagnostic laparoscopy or laparotomy
* Completion of preoperative systemic chemotherapy and preoperative laparoscopic HIPEC

Exclusion Criteria:

* Distant metastatic disease not limited to peritoneum: Solid organ metastases (liver, central nervous system, lung)
* Infections such as pneumonia or wound infections that would preclude protocol therapy
* Women with a positive urine or serum pregnancy test are excluded from this study; women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to refrain from breast feeding and practice adequate contraception as specified in the informed consent. Adequate contraception consists of oral contraceptive, implantable contraceptives, injectable contraceptives, a double barrier method, or abstinence
* Subjects with unstable angina or New York Heart Association grade II or greater congestive heart failure
* Subjects deemed unable to comply with study and/or follow-up procedures
* Subjects with a known hypersensitivity to protocol systemic chemotherapy that was life-threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Badgwell, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Badgwell B, Ikoma N, Murphy MB, Wang X, Estrella J, Roy-Chowdhuri S, Das P, Minsky BD, Lano E, Song S, Mansfield P, Ajani J. A Phase II Trial of Cytoreduction, Gastrectomy, and Hyperthermic Intraperitoneal Perfusion with Chemotherapy for Patients with Gastric Cancer and Carcinomatosis or Positive Cytology. Ann Surg Oncol. 2021 Jan;28(1):258-264. doi: 10.1245/s10434-020-08739-5. Epub 2020 Jun 17. PMID 32556731
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase II single arm trial at a single clinic and hospital from September 2016 to March 2019.
Pre-assignment Details: Exclusion criteria included stage IV disease outside of the peritoneum
Groups:
- Single Arm of Cytoreduction, Gastrectomy, and Intraperitoneal Chemotherapy: cytoreduciton, gastrectomy, and intraperitoneal chemotherapy
Period: Overall Study
Arm/Group | Single Arm of Cytoreduction, Gastrectomy, and Intraperitoneal Chemotherapy
Started | 20
Subtotal Gastrectomy | 11
Total Gastrectomy | 9
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm of Cytoreduction, Gastrectomy, and Intraperitoneal Chemotherapy
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: Years] | 58 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 20
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival from the date of diagnosis in subjects with stage IV gastric cancer
Time Frame: Date of diagnosis to date of death or last follow-up
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm of Cytoreduction, Gastrectomy, and Intraperitoneal Chemotherapy
Number analyzed (Participants) | 20
Months | 22.1 [15.4 to 30.3]

2. Secondary Outcome: Clavien-Dindo Surgical Complications
Description: 90-day surgical complications graded according to an accepted classification scale (Clavien-Dindo) Classification of Surgical Complications Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III: Requiring surgical, endoscopic or radiological intervention Grade IV: Life-threatening complication (including CNS complications)‡ requiring IC/ICU-management Grade V: Death of a patient
Time Frame: 90-days from surgery
Measure: Number; unit: events
Arm/Group | Single Arm of Cytoreduction, Gastrectomy, and Intraperitoneal Chemotherapy
Number analyzed (Participants) | 20
events
  Grade I and II | 15
  Grade III | 6
  Grade IV | 1

ADVERSE EVENTS:
Time Frame: Deaths were assessed up to 5 years. Complications according to the grading scale above were assessed 90 days from the date of surgery.
Description: We used the Clavien-Dindo surgical complication grading system, grade III and IV are considered major complications and perhaps similar to serious adverse events, of note, this system does not use the organ system classification of the CTCAE system
Groups:
- Cytoreduction, Gastrectomy, and Intraperitoneal Chemotherapy: Cytoreduction, Gastrectomy, and Intraperitoneal Chemotherapy
Arm/Group | Cytoreduction, Gastrectomy, and Intraperitoneal Chemotherapy
All-Cause Mortality (participants affected / at risk) | 14/20
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cytoreduction, Gastrectomy, and Intraperitoneal Chemotherapy (N=20)
Grade III (General disorders) | 6
Grade IV (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cytoreduction, Gastrectomy, and Intraperitoneal Chemotherapy (N=20)
Grade I (General disorders) | 1
Grade II (General disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT02891447/Prot_SAP_000.pdf